CLINICAL TRIAL: NCT05276401
Title: A Phase 2a, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Dose Escalating Study to Evaluate the Safety and Tolerability of Topically Applied Bisphosphocin Nu-3 Gel to Clinically Noninfected Chronic Diabetic Foot Ulcers (cDFU)
Brief Title: Nu-3 Topical Gel for Treatment of Diabetic Foot Ulcer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Request for additional preclinical data.
Sponsor: Lakewood-Amedex Inc (Industry)
Collaborators: Professional Education and Research Institute (Other); PrimeVigilance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LLA-Nu-3-CLIN002
Record Dates: First submitted 2022-02-25; First posted 2022-03-11 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-12

CONDITIONS: Chronic Diabetic Foot Ulcers
Keywords: Diabetic Foot; Metabolic Diseases; Skin Ulcer; Non-healing Wound; Diabetic Angiopathies; Foot Ulcer; Diabetic Neuropathies; Cardiovascular Diseases; Nu-3; Glucose Metabolism Disorders; DFU; Diabetes Mellitus; Endocrine System Diseases; Skin Diseases; Diabetes Complications; Non-healing Ulcer; Vascular Diseases; Leg Ulcer; Non-healing Wound Care; Bisphosphocin
MeSH Terms: conditions — Diabetic Foot; Metabolic Diseases; Skin Ulcer; Diabetic Angiopathies; Foot Ulcer; Diabetic Neuropathies; Cardiovascular Diseases; Glucose Metabolism Disorders; Diabetes Mellitus; Endocrine System Diseases; Skin Diseases; Diabetes Complications; Vascular Diseases; Leg Ulcer

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Dosage Form: Topical Antimicrobial Gel; Dosage: 5% Gel, 10% Gel; Frequency: BID for 28 days
  Interventions: Drug: 5% Bisphosphocin Topical Gel; Drug: 10% Bisphosphocin Topical Gel
- Placebo (Placebo Comparator): Dosage Form: Topical Gel; Dosage: Placebo; Frequency: BID for 28 days
  Interventions: Drug: Placebo Topical Gel

INTERVENTIONS:
Drug: 5% Bisphosphocin Topical Gel — Topical Gel
  Other Names: 5% Nu-3 Topical Gel
  Arms: Active
Drug: Placebo Topical Gel — Topical Gel
  Other Names: Placebo
  Arms: Placebo
Drug: 10% Bisphosphocin Topical Gel — Topical Gel
  Other Names: 10% Nu-3 Topical Gel
  Arms: Active

SUMMARY:
A PHASE 2a, MULTI-CENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED DOSE ESCALATING STUDY TO EVALUATE THE SAFETY AND TOLERABILITY OF TOPICALLY APPLIED BISPHOSPHOCIN NU-3 GEL TO CLINICALLY NONINFECTED CHRONIC DIABETIC FOOT ULCERS (cDFU)

DETAILED DESCRIPTION:
This is a Phase 2a, multi-center, randomized, double-blind, placebo-controlled, dose escalation study to evaluate the safety and tolerability of twice daily (BID) topically administered concentrations of Nu-3 gel in subjects with Type 1 and 2 diabetic non-healing target chronic diabetic foot ulcer (cDFU). The study will be conducted in 4 phases: Screening, SOC Run-In, Treatment, and a Safety Follow-up.

Subjects will have the study explained to them and will be provided the study specific informed consent form (ICF). For eligible subjects, the screening evaluations will be performed after the subject provides a written informed consent. For subjects enrolled in the study, activities will consist of two visits prior to randomization: screening visit, and a run-in visit; this will be followed by six scheduled visits (total = 8 visits). Screening will commence 14 days (± 2 days) prior to baseline visit.

During the screening period, a target cDFU will be established and characterized using information obtained from the subject's medical history. At the end of the screening and the beginning of the run-in SOC periods, subjects will have their selected target lesion assessed again. Those subjects whose target ulcers are shown to have ≥ 30% decrease in area will be considered as responders and will be discontinued from the study.

Non-responder subjects will enter the active treatment period and will be randomized in a 3:1 ratio into one of these dose cohorts in a dose escalating manner:

* Cohort 1: 5% Nu-3 gel + SOC (n = 12) or placebo gel + SOC (n = 4)
* Cohort 2: 10% Nu-3 gel + SOC (n = 12) or placebo gel + SOC (n = 4)

Study drug will be applied BID to the target cDFU for 28 days (± 2 days).

The decision to dose-escalate to the next higher concentration will be based on the recommendation of the Data Monitoring Committee (DMC) that will review all of the safety data from the previous subject cohort concurrent with the safety follow-up period. This decision will be based on pre-defined Dose Limiting Toxicity criteria (DLT), which will be detailed in the DMC charter. The maximum tolerated dose (MTD) will be considered as the dose level below that for which a DLT was observed. If the criteria for a DLT occurs in the initial dosing cohort then the study will be halted.

All randomized subjects will continue to receive SOC throughout the study per Appendix 4.

After completing the active treatment period, subjects will return after 2 weeks for a follow-up safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 18 years of age and up to 80 years of age, inclusive.
2. Voluntary written consent, given before performance of any clinical investigation-related procedure, and with the understanding that consent may be withdrawn at any time without prejudice to future medical care.
3. Non-hospitalized ambulatory subjects suffering from diabetes mellitus, Type I or II per ADA criteria.
4. The target ulcer is classified as grade 1 ulcer according to a Wagner Scale. These ulcers are superficial, full-thickness ulcers limited to the dermis, not extending to the subcutis.
5. Target ulcer is between 2 and 10 cm2 post debridement at screening and baseline.
6. The target ulcer must be no higher than the ankle (on or below the malleolus (ankle bone) with ≥50% below the malleolus.
7. Presence of a persistent cDFU for at least 4 weeks and not more than 1 year that has failed to respond to standard of care.
8. Adequate vascular perfusion as evidenced by one of the following:

   1. Dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 40 mmHg.
   2. Ankle Branchial Index (ABI) between 0.7 and 1.3 within 3 months of Screening using the extremity with the target ulcer.
   3. Arterial Doppler ultrasound evaluating for biphasic or triphasic dorsalis pedis and posterior tibial vessels at the level of the ankle or a TBI (Toe Brachial Index) of > 0.6 is acceptable.
9. Subject has a caregiver who is able to attend baseline visit and apply wound treatment and study dressings for the study duration.
10. Subject completed protocol-defined standardized wound care during the Screening and Run-in periods leading up to Day 0.
11. Must meet one of the following criteria:

    a. Female subjects of Non-Child-Bearing Potential defined as: i. Postmenopausal for at least 1 year, or surgically sterilized (i.e., hysterectomy or bilateral oophorectomy more than 3 months prior to Screening), or ii. Bilateral tubal ligation more than 6 months prior to Screening iii. Must have a negative serum β-hCG pregnancy test at screening and not be breastfeeding prior to being administered with the study drug.

    b. Male subjects of Non-Childbearing Potential defined as those vasectomized subjects whose vasectomy was performed 6 months prior to Screening or those diagnosed as sterile by a physician.

    c. Females and Males of Childbearing Potential who practice an acceptable method of contraception defined as the use of any form of hormonal contraceptive, a barrier method with spermicide, condoms, intrauterine device, or abstinence from sexual intercourse starting at least 60 days prior to Screening and continuing at least 30 days following the last treatment.
12. Subjects must be willing to undergo all clinical investigation-related procedures and attend all required visits.

Exclusion Criteria:

1. Ulceration with exposed tendon, capsule, or bone.
2. Suspicion of bone or joint infection by clinical or other criteria.
3. Unable or unwilling to utilize the standardized offloading RCW as required per protocol.
4. Target ulcer has decreased in area by ≥30% between Screening (V1) and Baseline (V3) visits.
5. Any subject that is currently on/requires oral, systemic or topical antibiotics, or is anticipated to require use during the course of the trial.
6. Any subject that has vascular compromise requiring surgical intervention or has undergone vascular reconstruction or angioplasty less than 1 month prior to randomization. Any planned surgical procedures during the study participation.
7. Serum Creatinine level >3.0 mg/dL.
8. Hemoglobin A1c (HbA1c) >12%.
9. Aspartate Aminotransferase (AST, GOT) and/or Alanine Aminotransferase (ALT, GPT) >3x the upper limit of normal.
10. Acute active Charcot foot.
11. The target ulcer is within 3 cm of any other ulcer.
12. Any subject that would be unable to safely monitor the infection status at home, and return for scheduled visits.
13. History of immunosuppression or taking immunosuppressive agents including systemic corticosteroids, except stable daily doses of 5 mg/day or less for chronic conditions.
14. Any subject with a life expectancy ≤ 6 months.
15. Pregnancy, including a positive pregnancy test at Screening or Baseline, or lactation.
16. Use of investigational drugs within 28 days prior to screening.
17. History of concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol.
18. Likely inability to comply with the protocol or cooperate fully with the investigator and site personnel.
19. Known or suspected active abuse of alcohol, narcotics, or non-prescription drugs.
20. Prior randomization in this clinical trial, or a previous Bisphosphocin study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumita Paul, MD, MPH, Study Director — Lakewood-Amedex Inc
Locations (5):
- United States (5):
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Limb Preservation Platform, Inc., Fresno, California
  - Doctors Research Network, South Miami, Florida
  - ACM Global Laboratories, Rochester, New York
  - Futuro Clinical Trials, LLC, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1: Active: Dosage Form: Topical Antimicrobial Gel; Dosage: 5%; Frequency: BID for 28 days
  Period 1: 5% Bisphosphocin Topical Gel: Topical Gel
- Period 1: Placebo: Dosage Form: Topical Gel; Dosage: Placebo; Frequency: BID for 28 days
  Period 1: Placebo Topical Gel: Topical Gel
- Period 2: Active: Dosage Form: Topical Antimicrobial Gel; Dosage: 10%; Frequency: BID for 28 days
  Period 2: 10% Bisphosphocin Topical Gel: Topical Gel
- Period 2: Placebo: Dosage Form: Topical Gel; Dosage: Placebo; Frequency: BID for 28 days
  Period 2: Placebo Topical Gel: Topical Gel
Period: Overall Study
Arm/Group | Period 1: Active | Period 1: Placebo | Period 2: Active | Period 2: Placebo
Started | 2 | 1 | 0 | 0
Completed | 2 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Number of Participants With Treatment-related Adverse Events After Nu-3 Gel Use on cDFU as Assessed by CTCAE v4.0
Description: Treatment emergent events related to clinical investigational product
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=2) | Placebo (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT05276401/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT05276401/SAP_002.pdf